CLINICAL TRIAL: NCT02081404
Title: Diagnosis of Acid Reflux Disease Using Novel Imaging: A Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Principal Investigator,, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: 3155105
Record Dates: First submitted 2012-04-06; First posted 2014-03-07 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Non-erosive Reflux Disease
Keywords: Non-erosive Reflux Disease
MeSH Terms: conditions — Non-Erosive Reflux Disease | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esomeprazole (Active Comparator): proton pump inhibitor
  Interventions: Drug: Esomeprazole
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — standard dose of proton pump inhibitor by mouth once a day for 30 days
  Other Names: Nexium
  Arms: Esomeprazole
Drug: Placebo — placebo
  Other Names: inactive substance
  Arms: Placebo

SUMMARY:
Gastroesophageal reflux disease (GERD), a common chronic disorder in the veteran population, is associated with drug costs exceeding $ 10 billion/year. Only 30-40% of patients with reflux symptoms have erosive esophagitis. The vast majority suffers from non erosive reflux disease (NERD), a condition in which standard endoscopy fails to identify any mucosal breaks and is unable to confirm the diagnosis. Unfortunately, a gold standard for the diagnosis of NERD does not exist. Narrow band imaging (NBI) utilizes spectral narrow band filters (incorporated into standard endoscopes) and helps to see abnormal areas not identified during standard endoscopy. Preliminary results have shown that NBI endoscopy may represent a significant improvement over standard endoscopy for the diagnosis of NERD. The purpose of this study is to accurately diagnosis non acid reflux disease by using a blue light (also known as NBI)upper endoscopy technique.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD), a common chronic disorder in the veteran population, is associated with drug costs exceeding $ 10 billion/year. Only 30-40% of patients with reflux symptoms have erosive esophagitis. The vast majority suffers from NERD; a condition in which standard endoscopy fails to identify any mucosal breaks and is unable to confirm the diagnosis. Unfortunately, a gold standard for the diagnosis of NERD does not exist. 24-hour esophageal pH monitoring and histologic esophageal mucosal changes in NERD patients have limited accuracy to be routinely used in clinical practice.

Narrow band imaging (NBI) utilizes spectral narrow band filters (incorporated into standard endoscopes) and enables imaging of features such as intrapapillary capillary loops (IPCLs); features not identified during standard endoscopy. Preliminary results have shown that NBI endoscopy may represent a significant improvement over standard endoscopy for the diagnosis of NERD. Our hypothesis is that NBI identifies changes in the distal esophagus that are specific for diagnosing patients with NERD. Specific Aim #1: To compare NBI features in the distal esophagus in patients with NERD (cases) and controls. Specific Aim #2: To determine whether the NBI features in NERD patients resolve after PPI therapy. Specific Aim #3: To correlate NBI findings with esophageal histology. Specific Aim #4: To assess the intra- and interobserver agreement for recognition of the proposed criteria for diagnosing NERD. Cases will be defined as patients with reflux symptoms (assessed by two validated questionnaires) with absent macroscopic erosions and abnormal esophageal pH results (NERD group). Control subjects will include patients with no reflux symptoms, absent macroscopic erosions and a normal esophageal pH result. To identify NBI findings as predictors of response, response to therapy in cases randomized to the PPI arm will be assessed using a validated GERD questionnaire and correlated with IPCL number and presence of microerosion. In addition, NBI findings in patients with reflux symptoms, no macroscopic erosions and normal esophageal pH result will also be compared with controls. Two biopsies will be obtained from the distal esophagus along with digital images and videorecordings.

Statistical analysis will be done as follows: Aim 1 - chi-square and t-test; with logistic regression and calculation of odds ratios, Aim 2- McNemar's test and kappa statistic, Aim 3- Spearman's correlation coefficient and Aim 4- intraclass correlation coefficient. Potential impact on Health Care: GERD is common among patients and by obviating the need for additional investigations and reducing unnecessary drug costs, NBI endoscopy could have a considerable positive impact on patients with NERD.

VA Project

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Capable of giving informed consents.
* Cases of NERD will be recruited on the basis of presence of heartburn and/or regurgitation using two validated GERD questionnaires in conjunction with an abnormal esophageal pH result and absence of erosions at standard endoscopy.
* Control subjects will include patients referred for an upper endoscopy for evaluation of non-reflux symptoms such as iron deficiency anemia, heme positive stools, screening of esophageal varices amongst others. A negative esophageal pH result and absence of erosions will be inclusion criteria for these patients.

Exclusion Criteria:

* Presence of macroscopic erosive esophagitis
* Pregnancy/lactation
* Chronic anticoagulation
* Patients with significant medical comorbidities (oxygen dependent chronic obstructive pulmonary disease, NYHA class III or IV congestive heart failure, recent diagnosis of cancer with a life-expectancy < 5 years)
* History of Barrett's esophagus
* Presence of columnar lined distal esophagus on endoscopy with intestinal metaplasia
* Presence of cancer or mass lesion in the esophagus or stomach
* Esophageal strictures
* Peptic ulcer disease and Helicobacter pylori infection
* Prior history of esophageal surgery
* Allergic to PPIs
* Patients on drugs known to cause pill-related esophagitis (e.g. potassium supplements)
* Patients with HIV or other immunocompromised conditions who may have infectious esophagitis
* Eosinophilic esophagitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
NBI endoscopy identifies changes in the distal esophagus that are specific for diagnosing patients with Non-Esophageal Reflux Disease. | 10 weeks
  1. Proportion of patients with NBI abnormalities in the NERD group vs. controls.
  2. Proportion of patients with resolution of NBI abnormalities after PPI therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, M.D., Principal Investigator — VA Office of Research and Development
Locations (2):
- Department of Veterans Affairs Medical Center, Kansas City, Missouri, United States
- Queen Medical Center, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participants individual participant data collected in the study will be available to other researchers upon request. Participants will be identified by participant number, age, race and gender. This information will be available at the end of the study and may be requested via email to april.higbee@va.gov.

REFERENCES:
- [Background] Sharma P, Wani S, Bansal A, Hall S, Puli S, Mathur S, Rastogi A. A feasibility trial of narrow band imaging endoscopy in patients with gastroesophageal reflux disease. Gastroenterology. 2007 Aug;133(2):454-64; quiz 674. doi: 10.1053/j.gastro.2007.06.006. Epub 2007 Jun 8. PMID 17681166
- [Background] Dent J, El-Serag HB, Wallander MA, Johansson S. Epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2005 May;54(5):710-7. doi: 10.1136/gut.2004.051821. PMID 15831922
- [Background] El-Serag HB. Time trends of gastroesophageal reflux disease: a systematic review. Clin Gastroenterol Hepatol. 2007 Jan;5(1):17-26. doi: 10.1016/j.cgh.2006.09.016. Epub 2006 Dec 4. PMID 17142109
- [Background] Liu JY, Woloshin S, Laycock WS, Rothstein RI, Finlayson SR, Schwartz LM. Symptoms and treatment burden of gastroesophageal reflux disease: validating the GERD assessment scales. Arch Intern Med. 2004 Oct 11;164(18):2058-64. doi: 10.1001/archinte.164.18.2058. PMID 15477443
- [Background] McDougall NI, Johnston BT, Kee F, Collins JS, McFarland RJ, Love AH. Natural history of reflux oesophagitis: a 10 year follow up of its effect on patient symptomatology and quality of life. Gut. 1996 Apr;38(4):481-6. doi: 10.1136/gut.38.4.481. PMID 8707073
- [Background] Talley NJ, Fullerton S, Junghard O, Wiklund I. Quality of life in patients with endoscopy-negative heartburn: reliability and sensitivity of disease-specific instruments. Am J Gastroenterol. 2001 Jul;96(7):1998-2004. doi: 10.1111/j.1572-0241.2001.03932.x. PMID 11467624
- [Background] Kulig M, Nocon M, Vieth M, Leodolter A, Jaspersen D, Labenz J, Meyer-Sabellek W, Stolte M, Lind T, Malfertheiner P, Willich SN. Risk factors of gastroesophageal reflux disease: methodology and first epidemiological results of the ProGERD study. J Clin Epidemiol. 2004 Jun;57(6):580-9. doi: 10.1016/j.jclinepi.2003.10.010. PMID 15246126
- [Background] Kulig M, Leodolter A, Vieth M, Schulte E, Jaspersen D, Labenz J, Lind T, Meyer-Sabellek W, Malfertheiner P, Stolte M, Willich SN. Quality of life in relation to symptoms in patients with gastro-oesophageal reflux disease-- an analysis based on the ProGERD initiative. Aliment Pharmacol Ther. 2003 Oct 15;18(8):767-76. doi: 10.1046/j.1365-2036.2003.01770.x. PMID 14535869
- [Background] Fass R, Ofman JJ. Gastroesophageal reflux disease--should we adopt a new conceptual framework? Am J Gastroenterol. 2002 Aug;97(8):1901-9. doi: 10.1111/j.1572-0241.2002.05912.x. PMID 12190152
- [Background] Fass R. Erosive esophagitis and nonerosive reflux disease (NERD): comparison of epidemiologic, physiologic, and therapeutic characteristics. J Clin Gastroenterol. 2007 Feb;41(2):131-7. doi: 10.1097/01.mcg.0000225631.07039.6d. PMID 17245209
- [Background] Carlsson R, Dent J, Watts R, Riley S, Sheikh R, Hatlebakk J, Haug K, de Groot G, van Oudvorst A, Dalvag A, Junghard O, Wiklund I. Gastro-oesophageal reflux disease in primary care: an international study of different treatment strategies with omeprazole. International GORD Study Group. Eur J Gastroenterol Hepatol. 1998 Feb;10(2):119-24. PMID 9581986
- [Background] Venables TL, Newland RD, Patel AC, Hole J, Copeman MB, Turbitt ML. Maintenance treatment for gastro-oesophageal reflux disease. A placebo-controlled evaluation of 10 milligrams omeprazole once daily in general practice. Scand J Gastroenterol. 1997 Jul;32(7):627-32. doi: 10.3109/00365529708996509. PMID 9246699
- [Background] Frazzoni M, De Micheli E, Savarino V. Different patterns of oesophageal acid exposure distinguish complicated reflux disease from either erosive reflux oesophagitis or non-erosive reflux disease. Aliment Pharmacol Ther. 2003 Dec;18(11-12):1091-8. doi: 10.1046/j.1365-2036.2003.01768.x. PMID 14653828
- [Background] Dent J, Brun J, Fendrick A, Fennerty M, Janssens J, Kahrilas P, Lauritsen K, Reynolds J, Shaw M, Talley N. An evidence-based appraisal of reflux disease management--the Genval Workshop Report. Gut. 1999 Apr;44 Suppl 2(Suppl 2):S1-16. doi: 10.1136/gut.44.2008.s1. No abstract available. PMID 10741335
- [Background] Dent J, Armstrong D, Delaney B, Moayyedi P, Talley NJ, Vakil N. Symptom evaluation in reflux disease: workshop background, processes, terminology, recommendations, and discussion outputs. Gut. 2004 May;53 Suppl 4(Suppl 4):iv1-24. doi: 10.1136/gut.2003.034272. PMID 15082609
- [Background] Kahrilas PJ, Quigley EM. Clinical esophageal pH recording: a technical review for practice guideline development. Gastroenterology. 1996 Jun;110(6):1982-96. doi: 10.1053/gast.1996.1101982. No abstract available. PMID 8964428
- [Background] Quigley EM. 24-h pH monitoring for gastroesophageal reflux disease: already standard but not yet gold? Am J Gastroenterol. 1992 Sep;87(9):1071-5. No abstract available. PMID 1519562
- [Background] Pandolfino JE, Lee TJ, Schreiner MA, Zhang Q, Roth MP, Kahrilas PJ. Comparison of esophageal acid exposure at 1 cm and 6 cm above the squamocolumnar junction using the Bravo pH monitoring system. Dis Esophagus. 2006;19(3):177-82. doi: 10.1111/j.1442-2050.2006.00561.x. PMID 16722995
- [Background] Pandolfino JE, Richter JE, Ours T, Guardino JM, Chapman J, Kahrilas PJ. Ambulatory esophageal pH monitoring using a wireless system. Am J Gastroenterol. 2003 Apr;98(4):740-9. doi: 10.1111/j.1572-0241.2003.07398.x. PMID 12738450
- [Background] Hirano I, Richter JE; Practice Parameters Committee of the American College of Gastroenterology. ACG practice guidelines: esophageal reflux testing. Am J Gastroenterol. 2007 Mar;102(3):668-85. doi: 10.1111/j.1572-0241.2006.00936.x. PMID 17335450
- [Background] Satoh K, Yamamoto H, Kawata H, Osawa H, Hanatsuka K, Kita H, Sunada K, Hirasawa T, Yoshizawa M, Ajibe H, Satoh Y, Sunada F, Sugano K. Comparison of hemostatic effects by route of H2 receptor antagonist administration following endoscopic mucosal resection in patients with neoplastic gastric lesions. Aliment Pharmacol Ther. 2005 Jun;21 Suppl 2:105-10. doi: 10.1111/j.1365-2036.2005.02483.x. PMID 15943856
- [Background] Lundell LR, Dent J, Bennett JR, Blum AL, Armstrong D, Galmiche JP, Johnson F, Hongo M, Richter JE, Spechler SJ, Tytgat GN, Wallin L. Endoscopic assessment of oesophagitis: clinical and functional correlates and further validation of the Los Angeles classification. Gut. 1999 Aug;45(2):172-80. doi: 10.1136/gut.45.2.172. PMID 10403727
- [Background] Amano Y, Ishimura N, Furuta K, Okita K, Masaharu M, Azumi T, Ose T, Koshino K, Ishihara S, Adachi K, Kinoshita Y. Interobserver agreement on classifying endoscopic diagnoses of nonerosive esophagitis. Endoscopy. 2006 Oct;38(10):1032-5. doi: 10.1055/s-2006-944778. PMID 17058170
- [Background] Kiesslich R, Kanzler S, Vieth M, Moehler M, Neidig J, Thanka Nadar BJ, Schilling D, Burg J, Nafe B, Neurath MF, Galle PR. Minimal change esophagitis: prospective comparison of endoscopic and histological markers between patients with non-erosive reflux disease and normal controls using magnifying endoscopy. Dig Dis. 2004;22(2):221-7. doi: 10.1159/000080323. PMID 15383765
- [Background] Yoshikawa I, Yamasaki M, Yamasaki T, Kume K, Otsuki M. Lugol chromoendoscopy as a diagnostic tool in so-called endoscopy-negative GERD. Gastrointest Endosc. 2005 Nov;62(5):698-703; quiz 752, 754. doi: 10.1016/j.gie.2005.06.027. PMID 16246682
- [Background] Numans ME, Lau J, de Wit NJ, Bonis PA. Short-term treatment with proton-pump inhibitors as a test for gastroesophageal reflux disease: a meta-analysis of diagnostic test characteristics. Ann Intern Med. 2004 Apr 6;140(7):518-27. doi: 10.7326/0003-4819-140-7-200404060-00011. PMID 15068979
- [Background] Dent J. Microscopic esophageal mucosal injury in nonerosive reflux disease. Clin Gastroenterol Hepatol. 2007 Jan;5(1):4-16. doi: 10.1016/j.cgh.2006.08.006. Epub 2006 Dec 8. PMID 17157563
- [Background] Tobey NA, Carson JL, Alkiek RA, Orlando RC. Dilated intercellular spaces: a morphological feature of acid reflux--damaged human esophageal epithelium. Gastroenterology. 1996 Nov;111(5):1200-5. doi: 10.1053/gast.1996.v111.pm8898633.
- [Background] Zentilin P, Savarino V, Mastracci L, Spaggiari P, Dulbecco P, Ceppa P, Savarino E, Parodi A, Mansi C, Fiocca R. Reassessment of the diagnostic value of histology in patients with GERD, using multiple biopsy sites and an appropriate control group. Am J Gastroenterol. 2005 Oct;100(10):2299-306. doi: 10.1111/j.1572-0241.2005.50209.x. PMID 16181384
- [Background] Gono K, Obi T, Yamaguchi M, Ohyama N, Machida H, Sano Y, Yoshida S, Hamamoto Y, Endo T. Appearance of enhanced tissue features in narrow-band endoscopic imaging. J Biomed Opt. 2004 May-Jun;9(3):568-77. doi: 10.1117/1.1695563. PMID 15189095
- [Background] Kumagai Y, Inoue H, Nagai K, Kawano T, Iwai T. Magnifying endoscopy, stereoscopic microscopy, and the microvascular architecture of superficial esophageal carcinoma. Endoscopy. 2002 May;34(5):369-75. doi: 10.1055/s-2002-25285. PMID 11972267
- [Background] el-Serag HB, Sonnenberg A. Associations between different forms of gastro-oesophageal reflux disease. Gut. 1997 Nov;41(5):594-9. doi: 10.1136/gut.41.5.594. PMID 9414963
- [Background] Sharma P, Bansal A, Mathur S, Wani S, Cherian R, McGregor D, Higbee A, Hall S, Weston A. The utility of a novel narrow band imaging endoscopy system in patients with Barrett's esophagus. Gastrointest Endosc. 2006 Aug;64(2):167-75. doi: 10.1016/j.gie.2005.10.044. PMID 16860063
- [Background] Abstracts of Digestive Disease Week, May 17-22, 2008 and the ASGE (American Society for Gastrointestinal Endoscopy) Postgraduate Course, May 21-22, 2008. San Diego, California, USA. Gastrointest Endosc. 2008 Apr;67(5):AB57-349. No abstract available. PMID 18578045
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology. 1997 May;112(5):1448-56. doi: 10.1016/s0016-5085(97)70025-8. PMID 9136821
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Risk factors associated with symptoms of gastroesophageal reflux. Am J Med. 1999 Jun;106(6):642-9. doi: 10.1016/s0002-9343(99)00121-7. PMID 10378622
- [Background] Locke GR, Talley NJ, Weaver AL, Zinsmeister AR. A new questionnaire for gastroesophageal reflux disease. Mayo Clin Proc. 1994 Jun;69(6):539-47. doi: 10.1016/s0025-6196(12)62245-9. PMID 8189759
- [Background] Shaw MJ, Talley NJ, Beebe TJ, Rockwood T, Carlsson R, Adlis S, Fendrick AM, Jones R, Dent J, Bytzer P. Initial validation of a diagnostic questionnaire for gastroesophageal reflux disease. Am J Gastroenterol. 2001 Jan;96(1):52-7. doi: 10.1111/j.1572-0241.2001.03451.x. PMID 11197287
- [Background] Fock KM, Teo EK, Ang TL, Tan JY, Law NM. The utility of narrow band imaging in improving the endoscopic diagnosis of gastroesophageal reflux disease. Clin Gastroenterol Hepatol. 2009 Jan;7(1):54-9. doi: 10.1016/j.cgh.2008.08.030. Epub 2008 Sep 3. PMID 18852068
- [Derived] Desai M, Srinivasan S, Sundaram S, Dasari C, Andraws N, Mathur S, Higbee A, Miller J, Beg S, Fateen W, Sami SS, Repici A, Ragunath K, Sharma P. Narrow-band imaging for the diagnosis of nonerosive reflux disease: an international, multicenter, randomized controlled trial. Gastrointest Endosc. 2022 Sep;96(3):457-466.e3. doi: 10.1016/j.gie.2022.04.020. Epub 2022 Apr 26. PMID 35487299